CLINICAL TRIAL: NCT04079972
Title: Personalized Lifestyle Intervention Based on SNP Testing and Weight Control
Brief Title: Personalized Lifestyle Intervention and Weight Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NaNa Keum (Other)
Collaborators: National Research Foundation of Korea (Other); DongGuk University (Other)
Responsible Party: Sponsor-Investigator, NaNa Keum, Associate Professor, DongGuk University
Organization: DongGuk University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018-12-006
Record Dates: First submitted 2019-02-18; First posted 2019-09-06 (Actual); Results first posted 2025-10-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-10

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Masking Description: This was an open-label randomized controlled trial; no masking was implemented for participants, investigators, or outcome assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Disclosure of obesity-related genetic risk with tailored lifestyle recommendations (Experimental): Participants received their obesity-related genetic test results, including variants in FTO (rs9939609), MC4R (rs17782313), and BDNF (rs6265), along with genotype-tailored lifestyle recommendations. The counseling materials encouraged risk-allele carriers to adopt healthier behaviors such as reducing fat intake, limiting snacking, and avoiding emotional eating. Personalized genetic results and recommendations were delivered at baseline through a user-friendly report.
  Interventions: Behavioral: Obesity-related genetic information disclosure with tailored lifestyle recommendations
- Disclosure of non-obesity-related genetic traits only (Active Comparator): Participants received genetic test results limited to non-obesity-related traits (e.g., beauty-related genes). They did not receive any obesity- or metabolism-related genetic information or tailored lifestyle recommendations. The full obesity-related genetic results were disclosed only after completion of the final follow-up.
  Interventions: Behavioral: Non-obesity-related genetic information disclosure

INTERVENTIONS:
Behavioral: Obesity-related genetic information disclosure with tailored lifestyle recommendations — They received their complete SNP results, including obesity-related traits, along with corresponding lifestyle recommendations.
  Arms: Disclosure of obesity-related genetic risk with tailored lifestyle recommendations
Behavioral: Non-obesity-related genetic information disclosure — Provided only with genetic test results related to beauty traits at baseline; information on metabolic health-related SNPs was disclosed only after the final follow-up assessment.
  Arms: Disclosure of non-obesity-related genetic traits only

SUMMARY:
This trial aims to investigate whether tailored lifestyle consultation through SNP testing leads to more effective weight loss among overweight or obese individuals compared to general lifestyle guidance for weight control.

ELIGIBILITY:
Inclusion Criteria:

1. Korean adults aged 18 years and older who are interested in weight management through dietary and/or exercise therapy.
2. Individuals who are able and willing to participate consistently for the entire 2-year study period.

Exclusion Criteria:

1. Individuals with any illness requiring regular medical treatment in a hospital.
2. Individuals currently taking long-term prescribed medications.
3. Individuals diagnosed with eating disorders or mental illnesses (e.g., depression, panic disorder) by a physician.
4. Individuals who have undergone gastric surgery for weight loss.
5. Individuals who have undergone heart surgery or cancer surgery.
6. Individuals with severe anemia.
7. Individuals who are unable to engage in physical exercise.
8. Pregnant or breastfeeding women, or those planning to become pregnant within 2 years.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2020-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: NaNa Keum, ScD, Principal Investigator — DongGuk University
Locations (1):
- Dongguk University, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Disclosure of Obesity-related Genetic Risk With Tailored Lifestyle Recommendations: Participants received their obesity-related genetic test results, including variants in FTO (rs9939609), MC4R (rs17782313), and BDNF (rs6265), along with genotype-tailored lifestyle recommendations. The counseling materials encouraged risk-allele carriers to adopt healthier behaviors such as reducing fat intake, limiting snacking, and avoiding emotional eating. Personalized genetic results and recommendations were delivered at baseline through a user-friendly report.
- Active Comparator: Disclosure of Non-Obesity-related Genetic Traits Only: Participants received genetic test results limited to non-obesity-related traits (e.g., beauty-related genes). They did not receive any obesity- or metabolism-related genetic information or tailored lifestyle recommendations. The full obesity-related genetic results were disclosed only after completion of the final follow-up.
Period: About 5 months after randomization
Arm/Group | Experimental: Disclosure of Obesity-related Genetic Risk With Tailored Lifestyle Recommendations | Active Comparator: Disclosure of Non-Obesity-related Genetic Traits Only
Started | 27 | 26
Completed | 20 | 21
Not Completed | 7 | 5
Period: About 17 months after randomization
Arm/Group | Experimental: Disclosure of Obesity-related Genetic Risk With Tailored Lifestyle Recommendations | Active Comparator: Disclosure of Non-Obesity-related Genetic Traits Only
Started | 20 | 21
Completed | 8 | 10
Not Completed | 12 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Disclosure of Obesity-related Genetic Risk With Tailored Lifestyle Recommendations | Active Comparator: Disclosure of Non-Obesity-related Genetic Traits Only | Total
Number analyzed (Participants) | 27 | 26 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 26 | 53
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.22 (2.80) | 22.31 (3.07) | 22.26 (2.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 16 | 16 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 27 | 26 | 53
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 27 | 26 | 53
Body Weight (kg) [Mean (Standard Deviation); unit: kg] | 74.3 (12.1) | 76.8 (11.2) | 75.6 (11.6)
Body fat mass (kg) [Mean (Standard Deviation); unit: kg] | 21.1 (9.8) | 23.1 (6.8) | 22.1 (8.4)
Body fat percentage (%) [Mean (Standard Deviation); unit: percentage] | 28.3 (10.7) | 31.1 (7.7) | 29.2 (9.3)
Skeletal muscle mass (kg) [Mean (Standard Deviation); unit: kg] | 29.8 (6.8) | 30.1 (6.0) | 29.9 (6.3)

OUTCOME MEASURES:

1. Primary Outcome: Body Weight (kg)
Description: Change was calculated as the value at the later time point minus the value at baseline (i.e., value at about 5 months after randomization minus baseline, and value at study completion (~17 months) minus baseline). Positive values represent increases from baseline, and negative values represent decreases.
Time Frame: About 5 months after randomization and at study completion (~17 months)
Population: number of started population differs from completed population
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Disclosure of obesity-related genetic risk with tailored lifestyle recommendations | Disclosure of non-obesity-related genetic traits only
Number analyzed (Participants) | 27 | 26
kg
  About 5 months after randomization: number analyzed (Participants) | 20 | 21
  About 5 months after randomization | 75.2 (13.2) | 79.2 (10.5)
  About 17 months after randomization: number analyzed (Participants) | 8 | 10
  About 17 months after randomization | 80.3 (19.4) | 74.5 (12.5)

2. Secondary Outcome: Body Fat Mass (kg)
Description: as for outcome 1
Time Frame: About 5 months after randomization and at study completion (~17 months)
Population: number of started population differs from completed population
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Disclosure of obesity-related genetic risk with tailored lifestyle recommendations | Disclosure of non-obesity-related genetic traits only
Number analyzed (Participants) | 27 | 26
kg
  About 5 months after randomization: number analyzed (Participants) | 20 | 21
  About 5 months after randomization | 21.4 (10.2) | 23.7 (7.0)
  About 17 months after randomization: number analyzed (Participants) | 8 | 10
  About 17 months after randomization | 25.9 (12.3) | 23.8 (8.0)

3. Secondary Outcome: Body Fat Percentage (%)
Description: as for outcome 1
Time Frame: About 5 months after randomization and at study completion (~17 months)
Population: number of started population differs from completed population
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Disclosure of obesity-related genetic risk with tailored lifestyle recommendations | Disclosure of non-obesity-related genetic traits only
Number analyzed (Participants) | 27 | 26
percentage
  About 5 months after randomization: number analyzed (Participants) | 20 | 21
  About 5 months after randomization | 28.5 (10.5) | 29.8 (7.8)
  About 17 months after randomization: number analyzed (Participants) | 8 | 10
  About 17 months after randomization | 31.8 (9.0) | 31.8 (8.4)

4. Secondary Outcome: Skeletal Muscle Mass (kg)
Description: as for outcome 1
Time Frame: About 5 months after randomization and at study completion (~17 months)
Population: number of started population differs from completed population
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Disclosure of obesity-related genetic risk with tailored lifestyle recommendations | Disclosure of non-obesity-related genetic traits only
Number analyzed (Participants) | 27 | 26
kg
  About 5 months after randomization: number analyzed (Participants) | 20 | 21
  About 5 months after randomization | 30.1 (7.1) | 31.1 (5.6)
  About 17 months after randomization: number analyzed (Participants) | 8 | 10
  About 17 months after randomization | 30.4 (7.4) | 28.1 (5.9)

ADVERSE EVENTS:
Time Frame: No adverse events were observed from enrollment through study completion (up to ~17 months).
Description: [Not Specified]
Arm/Group | Disclosure of Obesity-related Genetic Risk With Tailored Lifestyle Recommendations | Disclosure of Non-Obesity-related Genetic Traits Only
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/26
Other Adverse Events (participants affected / at risk) | 0/27 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-12-06): https://cdn.clinicaltrials.gov/large-docs/72/NCT04079972/Prot_002.pdf
  • Statistical Analysis Plan (2018-06-06): https://cdn.clinicaltrials.gov/large-docs/72/NCT04079972/SAP_003.pdf